CLINICAL TRIAL: NCT03258723
Title: Diabetes Prevention With Lifestyle Intervention and Metformin Escalation
Acronym: LIME
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 led to changes in study design and an early end to data collection.
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000020105; 1K12HL138037-01 (NIH); 1U54MD010711-01 (NIH)
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Patient Recruitment:
  The investigators are targeting the highest risk pre-diabetic patients for this study. Patient recruitment will occur through the involved health clinics.
  Control Participants Control participants in existing ECHORN sites (Puerto Rico, Barbados and Trinidad) will be recruited from the ECHORN Cohort Study (ECS).
  ECS does not have a recruitment site in New York; therefore, the New York LIME sites will need to recruit their own control participants, through random assignment of consented participants into the intervention and control groups. These participants will be offered a delayed intervention at the end of 2.5years, given the evidence supporting behavioral modification for diabetes prevention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Highest risk pre-diabetic patients
  Interventions: Behavioral: Lifestyle Intervention; Drug: Metformin
- Control (No Intervention): Control participants in existing ECHORN sites (Puerto Rico, Barbados and Trinidad) will be recruited. ECS does not have a recruitment site in New York; therefore, the New York LIME sites will need to recruit their own control participants, through random assignment of consented participants into the intervention and control groups.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The lifestyle intervention consists of a series of workshops adapted from the East Harlem Partnerships for Diabetes Prevention that discuss diabetes prevention, finding and affording healthy foods, label reading, physical activity, planning a healthy plate, making traditional foods healthy and portion control.
  The newly launched East Harlem Diabetes Prevention (EHDP) project's mobile app, iHEED will be used by intervention participants to help reinforce the content they learn during the workshop series.
  Arms: Intervention
Drug: Metformin — At 6 months, intervention participants who have not been able to lose weight or bring their HbA1c below the high risk range of 6% (determined by point-of-care testing) will have Metformin prescribed by their provider. Metformin will be prescribed at 500mg twice a day. If no change is seen at 12 months follow up, the dose will be increased to 850mg twice a day.
  Other Names: Glucophage
  Arms: Intervention

SUMMARY:
Specific Aim: Implement an evidence-based diabetes prevention pragmatic trial for high risk pre-diabetic individuals of Caribbean-descent to reduce the incidence of diabetes.

Hypothesis: This study seeks to test the hypothesis that implementation of a lifestyle intervention, with escalation to Metformin therapy will lower the incidence of diabetes among the highest risk pre-diabetic individuals of Caribbean-descent.

DETAILED DESCRIPTION:
The investigators propose to conduct a pragmatic trial that tests the effectiveness of lifestyle modification and Metformin use in minority populations. Our study population is Caribbean-descent individuals in Region 2, Trinidad and Barbados. The investigators will have five clinical intervention sites situated in New York - 2, Puerto Rico -1, Barbados -1, Trinidad -1 and US Virgin Islands -1. These sites were chosen because of the investigators' strong research network in these locations, and to enable us to address diabetes disparities due to geographic differences. The investigators will first modify an established lifestyle modification workshop series developed by the East Harlem Partnership for Diabetes Prevention (EHPDP) for use in the community, 10to target the population at the involved clinical sites. The investigators plan to adapt the D-CLIP protocol and escalate to Metformin therapy for the highest risk pre-diabetic patients whose hemoglobin A1c (HbA1c) has not improved or who remain morbidly obese.

The investigators will leverage our existing robust research infrastructure and network at the five sites through our Eastern Caribbean Health Outcomes Research Network (ECHORN) and now the Yale Transdisciplinary Collaborative center for Health Disparities focused on Precision Medicine (Yale-TCC). ECHORN is a research collaboration funded by the NIMHD (U2458849938) to address the burden of chronic disease in USVI, PR and the Eastern Caribbean. The Yale-TCC (U54MD010711) leverages the infrastructure and knowledge of the ECHORN, expands to include New York and New Jersey and focuses on diabetes and hypertension. The investigators' network includes community advisory boards as well as policy delegations that are well suited to inform this project and its expansion into routine healthcare practice and policy.

The control arm of this study was never activated due to COVID-19 restrictions.

ELIGIBILITY:
Inclusion Criteria:

* BMI>25 or WC>88/102cm
* No history of type I or type II diabetes or gestational diabetes
* Not on blood sugar altering medication
* Ability to attend weekly sessions
* HbA1c 6-6.4%

Exclusion Criteria:

* Pregnant
* eGFR<45 mL/min/1.73 m2
* Prescribed Metformin and randomized to the control arm

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Nunez-Smith, MD, Principal Investigator — Yale University
Locations (4):
- University of the West Indies, Cavehill and Barbados Ministry of Health Polyclinics, Bridgetown, Barbados
- Internal Medicine Clinic at the University of Puerto Rico Hospital, Carolina, Puerto Rico
- Southwest Regional Health Authority, La Romaine Health Center, San Fernando, Trinidad and Tobago
- Ministry of Health Clinics, Charlotte Amalie, Virgin Islands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassan S, Sobers NP, Paul-Charles J, Herbert J, Dharamraj K, Galusha D, Cruz E, Garcia-Rivera E, Fredericks L, Arniella G, Cattamanchi A, Adams OP, Maharaj RG, Nazario CM, Nunez M, Nunez-Smith M. Diabetes prevention in the Caribbean using lifestyle intervention and Metformin escalation (LIME): results from a quasi-experimental study. BMC Public Health. 2025 Nov 22;25(1):4409. doi: 10.1186/s12889-025-25291-7. PMID 41275221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 211 participants agreed to be a part of the study, 114 participants attended at least 1 workshop and are those considered "enrolled".
Groups:
- Intervention: Highest risk pre-diabetic patients
  Lifestyle Intervention: The lifestyle intervention consists of a series of workshops adapted from the East Harlem Partnerships for Diabetes Prevention that discuss diabetes prevention, finding and affording healthy foods, label reading, physical activity, planning a healthy plate, making traditional foods healthy and portion control.
  The newly launched East Harlem Diabetes Prevention (EHDP) project's mobile app, iHEED will be used by intervention participants to help reinforce the content they learn during the workshop series.
  Metformin: At 6 months, intervention participants who have not been able to lose weight or bring their HbA1c below the high risk range of 6% (determined by point-of-care testing) will have Metformin prescribed by their provider. Metformin will be prescribed at 500mg twice a day. If no change is seen at 12 months follow up, the dose will be increased to 850mg twice a day.
Period: Overall Study
Arm/Group | Intervention
Started | 114
6 Month Follow up | 80
12 Month Follow up | 52
Completed | 52
Not Completed | 62
Not completed — COVID Interruption of study | 54
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 1
  Race/Ethnicity: Black or African or Caribbean | 67
  Race/Ethnicity: Asian | 26
  Race/Ethnicity: Hispanic or Latino or Puerto Rican | 1
  Race/Ethnicity: Mixed or multi-racial | 18
  Race/Ethnicity: Unknown/Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 114
Education [Count of Participants; unit: Participants] — Population: 1 participant missing education information.
  Participants
    number analyzed (Participants) | 113
    Less than high school | 14
    High school | 45
    Some college | 28
    College or more | 26
HbA1c [Mean (Standard Deviation); unit: percentage] | 6.2 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c)
Description: Hemoglobin A1C (HbA1C) test was assessed via clinical tests.
Time Frame: Baseline and 12 months
Population: All participants with valid data on matched cases at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Intervention
Number analyzed (Participants) | 51
percentage
  Baseline | 6.19 (0.15)
  12 Months | 5.67 (0.50)
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Change in Weight (kg)
Description: Weight in kilograms (kg) assessed via clinical tests.
Time Frame: Baseline and 6 months
Population: Participants with valid data that could be matched from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention
Number analyzed (Participants) | 76
kg
  Baseline | 86.66 (16.63)
  6 Months | 85.00 (16.86)
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases; Test type: Superiority; p = 0.0005, t-test, 2 sided

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure assessed via clinical tests.
Time Frame: Baseline and 6 months
Population: Participants with valid data matched from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 74
mmHg
  Baseline | 133.93 (20.72)
  6 Months | 131.64 (18.54)
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases; Test type: Superiority; p = 0.1809, t-test, 2 sided

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure assessed via clinical tests.
Time Frame: Baseline and 6 months
Population: Participants with valid data matched from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 74
mmHg
  Baseline | 84.86 (11.87)
  6 Months | 82.54 (10.49)
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases; Test type: Superiority; p = 0.0973, t-test, 2 sided

5. Secondary Outcome: Diabetes Risk Score
Description: The Diabetes Risk Score has been designed to be a screening tool for identifying high-risk subjects in the population and for increasing awareness of the modifiable risk factors and healthy lifestyle. The score ranges from 0-20, with a higher score indicating higher risk.
Time Frame: 6 months
Population: These data were not collected.
Arm/Group | Intervention
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Self-Efficacy Score - Personal Control Scale
Description: The Self-efficacy survey is an excerpt from the 43-item Risk Perception Survey for Developing Diabetes, designed for people at high risk for developing diabetes. It measures perceived comparative and environmental risk for developing diabetes. Scoring for the self-efficacy questions is done by an average and ranges from 1 to 4, with a higher score indicating more perceived risk.
Time Frame: Baseline and 6 months
Population: Matched cases with valid data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 68
units on a scale
  Baseline | 3.55 (0.50)
  6 Months | 3.64 (0.43)
Statistical Analysis 1: Comparison: Intervention; Within subject change on matched cases; Test type: Superiority; p = 0.1992, t-test, 2 sided

7. Secondary Outcome: Change in Self-Efficacy Score - Worry Scale
Description: as for outcome 6
Time Frame: 6 months
Population: Matched cases with valid data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 68
units on a scale
  Baseline | 2.88 (1.01)
  6 Months | 2.83 (0.94)
Statistical Analysis 1: Comparison: Intervention; Within subject change on matched cases; Test type: Superiority; p = 0.7017, t-test, 2 sided

8. Secondary Outcome: Change in Physical Activity Level.
Description: Change in physical activity level was assessed using the self-reported WHO Physical Activity Questionnaire
Time Frame: Baseline and 6 months
Population: Participants with valid data that could be matched from baseline to 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 70
Participants
  Baseline: Low | 22
  Baseline: Moderate | 22
  Baseline: High | 26
  6 Months: Low | 28
  6 Months: Moderate | 18
  6 Months: High | 24
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases in low activity group at baseline; Test type: Superiority; p = 0.1573, McNemar
Statistical Analysis 2: Comparison: Intervention; Within group change from baseline assessed on matched cases in medium activity group at baseline; Test type: Superiority; p = 0.4328, McNemar
Statistical Analysis 3: Comparison: Intervention; Within group change from baseline assessed on matched cases in high activity group at baseline; Test type: Superiority; p = 0.6698, McNemar

9. Secondary Outcome: Change in Fruit and Vegetable Intake (Total Servings)
Description: Total mean servings per day of fruit and vegetables self report via electronic survey.
Time Frame: Baseline and 6 months
Population: Participants with valid data that could be matched from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: daily servings
Arm/Group | Intervention
Number analyzed (Participants) | 70
daily servings
  Baseline | 1.53 (0.97)
  6 Months | 1.61 (1.02)
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases; Test type: Superiority; p = 0.5271, t-test, 2 sided

10. Secondary Outcome: Change in Sugar-sweetened Beverage Intake (Teaspoons Per Day)
Description: Change in mean teaspoons per day of sugar-sweetened beverage intake self report via electronic survey.
Time Frame: Baseline and 6 months
Population: Participants with valid data that could be matched from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: teaspoons
Arm/Group | Intervention
Number analyzed (Participants) | 68
teaspoons
  Baseline | 7.30 (8.08)
  6 Months | 3.83 (4.10)
Statistical Analysis 1: Comparison: Intervention; Within group change from baseline assessed on matched cases; Test type: Superiority; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT03258723/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT03258723/SAP_001.pdf
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03258723/ICF_002.pdf